CLINICAL TRIAL: NCT00642655
Title: A Phase I/II Trial to Investigate the Safety and Efficacy of Rituximab and IVIG as Agents to Desensitize Highly-HLA Sensitized Dialysis Patients Awaiting Kidney Transplantation
Brief Title: Rituximab and Intravenous Immunoglobulin (IVIG) for Desensitization in Renal Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Genentech, Inc. (Industry); Biogen (Industry)
Responsible Party: Stanley C. Jordan, MD, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U3176s
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Kidney Transplant
Keywords: IVIG; Rituximab; Highly Sensitized; Kidney Transplantation
MeSH Terms: interventions — Immunoglobulins, Intravenous; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IVIG and Rituximab — IVIG 2gm/kg given intravenously on day#0 and day#30 Rituximab 1gm given intravenously on day#7 and day#22

SUMMARY:
The purpose of this study is to examine the safety and efficacy of IVIG in combination with Rituximab to lower the level of HLA-sensitive antibodies and block their ability to attack a transplanted organ in patients who are highly HLA-sensitized and are awaiting transplantation.

DETAILED DESCRIPTION:
Patients eligible for the study will be those who have anti-HLA antibody (Panel Reactive Antibody {PRA}) of >30%. If patients meet these criteria, patients will be asked to have an assessment of the ability of IVIG to reduce the anti-HLA antibodies activity in the test tube. Patients will receive IVIG 2gm/kg x1 on hemodialysis. Seven days later, patients will receive Rituximab 1gm in the CSMC Infusion Center as per protocol for Rituximab infusion. The second Rituximab infusion will be on day #22. Additional IVIG infusion will be given at month one.

Patients will continue to be followed for an additional 12 months after the last IVIG infusion and will be asked to return for follow up visits at month 1 through 5, month 7 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the study will be those who have anti-HLA antibody (Panel Reactive Antibody [PRA]) of >30% and are eligible for transplantation at Cedars-Sinai Medical Center. We currently anticipate entering 20 patients over the course of the study. We currently have ~100 patients on our wait list that would meet the above criteria. Patients will be selected based on the ability of IVIG to inhibit the cytotoxic anti-HLA antibody activity in vitro. They will then receive IVIG 2gm/kg X1 on day 1 while on hemodialysis. Seven days later, the patients will receive Rituxan® 1gm in the CSMC Cancer Infusion Center as per protocol for Rituxan® infusion. The second Rituxan® infusion will be on day#22. The patients will have monitoring of anti-HLA antibody and outlined tests as shown above.
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Adequate liver function, as indicated by normal liver function tests (NL: AST, ALT, Bilirubin and negative tests for hepatitis C and hepatitis B.
* Negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.

Exclusion Criteria:

* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)

  * Receipt of a live vaccine within 4 weeks prior to randomization
  * Previous Treatment with Rituximab (MabThera® / Rituxan®)
  * Prior antibody therapy
  * History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
  * History of HIV (positive HIV, HIV conducted during screening)
  * History of Hepatitis B and/or Hepatitis C
  * History of recurrent significant infection or history of recurrent bacterial infections
  * Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
  * Lack of peripheral venous access
  * History of drug, alcohol, or chemical abuse within 6 months prior to screening
  * Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or lactation
  * Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
  * History of psychiatric disorder
  * Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
  * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
  * Inability to comply with study and follow-up procedures

Laboratory Exclusion Criteria (at Screening)

* Hemoglobin: < 8.5 gm/dL
* Platelets: < 100,000/mm
* AST or ALT >2.5 x Upper Limit of Normal unless related to primary disease.
* Positive Hepatitis B or C serology
* Positive HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Success of transplantation | 12 months

SECONDARY OUTCOMES:
Number and severity of rejection episodes | 12

CONTACTS AND LOCATIONS:
Overall Officials: Stanley C. Jordan, MD, Principal Investigator — Cedars-Sinai Medical Center; Ashley A Vo, PharmD, Study Director — Cedars-Sinai Medical Center
Locations (1):
- 8700 Beverly Blvd., Los Angeles, California, United States

REFERENCES:
- [Derived] Vo AA, Lukovsky M, Toyoda M, Wang J, Reinsmoen NL, Lai CH, Peng A, Villicana R, Jordan SC. Rituximab and intravenous immune globulin for desensitization during renal transplantation. N Engl J Med. 2008 Jul 17;359(3):242-51. doi: 10.1056/NEJMoa0707894. PMID 18635429